CLINICAL TRIAL: NCT06877377
Title: A Pilot Randomized, Blinded, Placebo-controlled Study of the Safety and Efficacy of Natural Genome Reconstruction Technology of Hematopoietic Stem Cells in Adult Patients
Brief Title: Study of the Safety and Efficacy of Natural Genome Reconstruction Technology of Hematopoietic Stem Cells in Adult Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center for New Medical Technologies, Novosibirsk, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SW025
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Aging
Keywords: DNAgr-technology; haemopoesis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: hDNAgr Technology (Experimental): Participants in this arm will receive the hDNAgr therapy, a novel approach using fragmented double-stranded DNA designed to correct damaged genomic regions in hematopoietic stem cells and elongate telomeres. The treatment is administered according to the protocol schedule (Visits at Day 0, 14, 28, 60, 90, and 180), and all relevant safety and efficacy parameters (adverse events, hematological markers, telomere length, and potential aging biomarkers) are assessed throughout the 6-month follow-up period.
  Interventions: Biological: hDNAgr Therapy
- Placebo Comparator: Inactive Formulation (Placebo Comparator): Participants in this arm will receive an inactive placebo formulation, identical in appearance to the hDNAgr therapy but lacking the active DNA fragments. This ensures blinding for both subjects and investigators. The same follow-up schedule (Visits at Day 0, 14, 28, 60, 90, and 180) and assessments (adverse events, hematological markers, telomere length, and aging biomarkers) are conducted, enabling direct comparison to the experimental arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: hDNAgr Therapy — A novel investigational therapy that uses fragmented therapeutic double-stranded DNA, designed to correct or replace locally damaged genomic regions in hematopoietic stem cells and elongate telomeres. The hDNAgr therapy is administered according to the study protocol schedule (Visits at Day 0, 14, 28, 60, 90, and 180), with blood draws and safety evaluations at each time point to assess hematological parameters, telomere length, and potential impacts on biological aging.
  Arms: Experimental: hDNAgr Technology
Other: Placebo — An inactive formulation identical in appearance to the hDNAgr therapy but lacking the active DNA fragments. It is administered under the same schedule and conditions as the experimental intervention to maintain blinding and enable comparison of safety and efficacy outcomes.
  Arms: Placebo Comparator: Inactive Formulation

SUMMARY:
This pilot randomized, double-blind, placebo-controlled study evaluates the safety and efficacy of the hDNAgr technology aimed at natural genome reconstruction in hematopoietic stem cells in adults aged 45-65. The study hypothesizes that administering fragmented therapeutic double-stranded DNA will safely correct localized genomic damage-including telomere elongation-enhance hematopoietic function by restoring polyclonality and increasing reparative potential, and ultimately rejuvenate blood and bone marrow to potentially lower the patient's biological age. The primary endpoint is safety and tolerability, assessed by the frequency and severity of adverse events, while secondary endpoints focus on telomere length, hematological parameters, aging and inflammation biomarkers, functional health measures, and preliminary biological age evaluations. Sixty participants (30 in the hDNAgr group and 30 receiving placebo) will be observed over a 6-month period with multiple scheduled visits.

DETAILED DESCRIPTION:
This pilot study, titled "Pilot Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Natural Genome Reconstruction Technology in Hematopoietic Stem Cells in Adult Patients," investigates the use of hDNAgr technology-which involves the administration of fragmented therapeutic double-stranded DNA-to achieve natural genomic reconstruction in hematopoietic stem cells. The hypothesis is that this intervention will lead to a safe and controlled correction of damaged genomic regions and telomere elongation, thereby improving hematopoietic parameters (evidenced by restored polyclonality and enhanced reparative potential) and promoting overall rejuvenation of the blood and bone marrow, with the potential to reduce the patient's biological age. The primary endpoint is the safety and tolerability of the therapy, determined by the incidence and severity of adverse events (AEs) and serious adverse events (SAEs) over the study period. Secondary endpoints include changes in telomere length (using methods like Q-FISH or qPCR), detailed hematological assessments (hemoglobin levels, counts of erythrocytes, leukocytes, platelets, differential leukocyte analysis, and CD34⁺ cell counts), evaluation of biomarkers of aging and systemic inflammation (such as IL-6, CRP, and TNF-α), functional health assessments (e.g., via the SF-36 scale), and preliminary measures of biological age (including epigenetic clocks). Eligible participants are men and women aged 45-65 who have no decompensated chronic diseases, no history of malignancies in the past 5 years, and who provide informed consent and adhere to study protocols. Exclusion criteria include pregnancy, lactation, plans for pregnancy during the study, active immune deficiencies, decompensated cardiovascular/hepatic/renal conditions, recent use of immunosuppressive or chemotherapeutic agents, substance dependency, and participation in other clinical trials within 30 days of enrollment. The study protocol includes an initial screening (Visit 0), baseline randomization and measurements (Visit 1, Day 0), interim visits at approximately Days 14, 28, 60, and 90, and a final evaluation at Day 180. With 60 participants randomized equally between the hDNAgr and placebo groups, this 6-month pilot trial is designed to generate primary data on safety, tolerability, and preliminary efficacy, thereby setting the stage for future phase II/III studies and potential expansion of indications.

ELIGIBILITY:
Inclusion Criteria:

* . Men and women aged 45 to 65 years inclusive (optimal age range for a pilot study of the effect on aging processes).
* Confirmed absence of serious chronic diseases in the decompensation stage (based on the results of a standard clinical and laboratory examination).
* No history of malignant neoplasms over the past 5 years. Written informed consent to participate in the study. Willingness to comply with the study protocol, including attending all scheduled visits and undergoing the required diagnostic procedures.

Exclusion Criteria:

* Pregnancy, lactation, or planning a pregnancy during the study.
* The presence of immunodeficiency states (HIV infection, severe autoimmune diseases, etc.) in the acute stage.
* Decompensated cardiovascular, hepatic, renal pathologies (a conclusion from a therapist or a specialized specialist is required).
* Take immunosuppressants, corticosteroids or chemotherapeutic drugs within 3 months before screening.
* Alcohol or drug addiction, confirmed by medical documents or identified during screening.
* Participation in other clinical trials 30 days before inclusion or planned participation during this study.
* Observation plan, duration of Follow-Up and number of visits

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Any Treatment-Emergent Adverse Events (Safety and Tolerability) in Male Participants Receiving hDNAgr Therapy | 180 days
  The primary endpoint is the frequency and severity of adverse events (AEs) and serious adverse events (SAEs) observed in participants receiving hDNAgr therapy versus placebo. Safety will be assessed at each study visit through medical examinations, laboratory evaluations, and participant-reported outcomes.

SECONDARY OUTCOMES:
Change in Telomere Length | 180 days
  Telomere length in peripheral blood leukocytes will be measured using validated methods (e.g., Q-FISH, qPCR) to assess potential elongation or maintenance over time.
Hemoglobin Level (g/dL) | 180 days
  Hemoglobin concentration (g/dL) measured in peripheral blood. Values will be obtained via standard clinical laboratory methods to assess potential improvements or changes in oxygen-carrying capacity.
Red Blood Cell (RBC) Count (×10^12/L) | 180 days
  RBC count (×10^12 per liter) measured in peripheral blood using automated counters to evaluate overall erythropoietic activity and red cell status.
White Blood Cell (WBC) Count (×10^9/L) | 180 days
  WBC count (×10^9 per liter) in peripheral blood determined by automated hematology analyzers to monitor immune cell populations and potential shifts in leukocyte levels.
WBC Differential (%) | 180 days
  Distribution percentages of neutrophils, lymphocytes, monocytes, eosinophils, and basophils in peripheral blood. This measure helps to evaluate shifts in immune cell subtypes over time.
Platelet Count (×10^9/L) | 180 days
  Platelet count (×10^9 per liter) measured in peripheral blood with an automated analyzer. This outcome assesses platelet production and turnover.
CD34⁺ Hematopoietic Stem Cell Count (cells/µL) | 180 days
  Absolute count of CD34⁺ progenitor cells (cells/µL) in peripheral blood, typically assessed via flow cytometry. Helps gauge changes in hematopoietic stem cell populations over the course of therapy.
Preliminary Biological Age Evaluation | 180 days
  Assessment of biological age via methods such as epigenetic clocks and/or relevant functional tests to gauge any potential "rejuvenation" effect of the therapy.
36-Item Short Form Health Survey (SF-36) Score | 180 days
  The SF-36 (Short Form Health Survey) is a 36-item validated questionnaire assessing eight domains of physical and mental health: Physical Functioning, Role Limitations due to Physical Health, Bodily Pain, General Health, Vitality, Social Functioning, Role Limitations due to Emotional Problems, and Mental Health. Scores for each domain range from 0 to 100, with higher scores indicating better perceived health status. Composite scores (Physical Component Summary and Mental Component Summary) are also reported on a 0-100 scale, where 0 represents the poorest health and 100 represents the best health.
Interleukin-6 (IL-6) Level (pg/mL) | 180 days
  Serum IL-6 concentrations will be measured in picograms per milliliter (pg/mL) using a validated immunoassay to evaluate changes in systemic inflammation over time. Higher levels may indicate increased inflammatory activity.
C-Reactive Protein (CRP) Level (mg/L) | 180 days
  CRP will be measured in milligrams per liter (mg/L) to assess the presence and degree of systemic inflammation, with higher levels indicating a more pronounced inflammatory state.
Tumor Necrosis Factor Alpha (TNF-α) Level (pg/mL) | 180 days
  TNF-α will be measured in picograms per milliliter (pg/mL) via a validated immunoassay to evaluate changes in systemic inflammatory and immune responses over time.

IPD SHARING:
Plan to Share IPD: No